CLINICAL TRIAL: NCT00272597
Title: Risperidone Long Acting: A Healthcare Resource Utilization Pilot Study
Brief Title: Risperidone LA Heathcare Resource Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Riverview Hospital (Unknown)
Responsible Party: Principal Investigator, Ric Procyshyn, Principle Investigator, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C05-0356
Record Dates: First submitted 2006-01-03; First posted 2006-01-06 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Psychosis; Schizophrenia
Keywords: Psychosis; schizophrenia; schizoaffective; risperidone
MeSH Terms: conditions — Psychotic Disorders; Schizophrenia | interventions — Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Risperidone LAI (Other): Subjects treated with any antipsychotic can be switched to Risperidone LAI.
  * If the subject is currently treated with an antipsychotic other than risperidone, the dosage will be tapered gradually and discontinued. Simultaneously, oral risperidone will be started at 2 mg/day and increased to no more than 6 mg/day. The subject will be treated with risperidone monotherapy for at least five days prior to entering the stabilization phase of the study.
  * On the other hand, if the patient has already been treated for more than 5 days with risperidone monotherapy then he/she may enter the stabilization phase of the study immediately.
  Interventions: Drug: Risperidone

INTERVENTIONS:
Drug: Risperidone — See Detailed Description.

SUMMARY:
The primary objective of this pilot study is to evaluate the impact of switching 30 subjects from an existing antipsychotic to risperidone long acting on healthcare resource utilization. The study will be a ten month open-label, 'mirror-image', pilot study. Healthcare resource utilization during the 10 months prior to starting risperidone long acting will be retrospectively collected for all subjects (period A) at the beginning of the study. The utilization of direct medical resources will also be collected for 10 months after initiation of risperidone long acting (period B). In this design the patients will serve as their own control.

DETAILED DESCRIPTION:
Screening (Week -2 to Week 0; Days -14 to -1) In this phase, the subject is required to be treated with oral risperidone (as their only antipsychotic) for a period of at least 5 days before entering the stabilization phase of the study. Therefore,

* If the subject is currently treated with an antipsychotic other than risperidone, the dosage will be tapered gradually and discontinued. Simultaneously, oral risperidone will be started at 2 mg/day and increased to no more than 6 mg/day. The subject will be treated with risperidone monotherapy for at least five days prior to entering the stabilization phase of the study.
* On the other hand, if the patient has already been treated for more than 5 days with risperidone monotherapy then he/she may enter the stabilization phase of the study immediately.

Stabilization Phase (Weeks 1 - 14; Days 0 - 98) The first three doses of risperidone long acting (Days 0, 14 and 28) will be 25 mg for all subjects. At the time of the fourth injection (Day 42), the dosage of risperidone long acting may be increased from 25 mg IM to 37.5 mg IM upon discretion of the treating physician. Further increases in the dosage of risperidone long acting may be made at the time of the 6th and 8th injections (Days 70 and 98 respectively). In this case, if the subject is currently receiving 25 mg he/she may be increased to 37.5 mg but not 50 mg. Alternatively, if the patient is currently receiving 37.5 mg, then subject may be increased to the maximum recommended dosage of 50 mg IM every two weeks.

To accommodate for the latency period (i.e., the time for risperidone to be released from the microspheres and approach therapeutic plasma levels), subjects entering into the study will continue on oral risperidone for the first three weeks (Days 0-21). Temporary oral supplementation will also be permitted anytime during the stabilization phase of the study when considered by the treating physician to be clinically necessary for the treatment of breakthrough psychosis. With only one exception, the treating physician is not restricted from adding or discontinuing any pharmacological treatment deemed necessary for the clinical management of the subject. The exception in this case prohibits the addition of another antipsychotic agent and applies only to the stabilization phase of the study.

Maintenance Phase (Weeks 15 - 38; Days 99 - 266) Patients that have shown adequate response to risperidone long acting will continue into the maintenance phase of the study. From this point onwards, the treating physician may change the dosage of risperidone long acting at any time as considered necessary. Temporary oral supplementation will also be permitted during the maintenance phase when considered by the treating physician to be clinically necessary for the treatment of breakthrough psychosis. Apart from the above, the treating physician is not restricted from adding or discontinuing any pharmacological treatment (including another antipsychotic) deemed necessary for the clinical management of the subject.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a diagnosis of schizophrenia or schizoaffective disorder according to DSM-IV criteria.
* Men and women, aged 18-65 years.
* Subjects must be able to give written informed consent.
* Subjects must be inpatients.
* Subjects must have adequate data to assess healthcare resource utilization for the previous 10 months.
* Subjects must have been previously treated with (and tolerated) oral risperidone.
* Results of standard clinical laboratory tests are to be within the laboratory's reference range or, if outside this range, judged by the investigator to be not clinically significant.

Exclusion Criteria:

Exclusion Criteria:

* Subjects with significant alcohol or substance abuse in the past 3 months.
* Subjects with other psychiatric, medical or behavioural comorbid disorder that in the opinion of the investigator may interfere with study conduct or interpretation (such as delirium, stroke, developmental disability).
* Subjects who are pregnant, breast-feeding, or women of child-bearing potential not using adequate contraception.
* Subjects with known hypersensitivity or allergy to risperidone.
* Subjects with tardive dyskinesia or a history of neuroleptic malignant syndrome.
* Subjects with a known history of being unresponsive to risperidone.
* Subjects with a clinically significant electrocardiogram abnormality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-09; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To assess the impact of switching subjects from an existing antipsychotic to risperidone long acting on healthcare resource utilization. This will be evaluated by assessing:
Direct cost of care
Frequency and duration of institutional care
Discharge
Relapse

SECONDARY OUTCOMES:
To determine if effectiveness is maintained for subjects switched from an existing antipsychotic to risperidone long acting. This will be evaluated by assessing:
Positive and negative symptoms (PANSS)
Overall illness severity (CGI severity, CGI improvement)
Social and occupational functioning (SOFAS), and
Remission
To evaluate the safety and tolerability of risperidone long acting. This will be evaluated by assessing:
Extrapyramidal symptoms (ESRS)
Side effects (UKU side effect rating scale)
Akathisia (Barnes akathisia scale)
Quality of life (SF-36)
Weight, and waist circumference
Hematology (fasting glucose and lipid analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Ric Procyshyn, MD, Principal Investigator — The University of British Columbia
Locations (1):
- Riverview Hospital, Coquitlam, British Columbia, Canada

REFERENCES:
- [Derived] Procyshyn RM, Barr AM, Flynn S, Schenk C, Ganesan S, Honer WG. Long-acting injectable risperidone in treatment refractory patients: a 14-week open-label pilot study. Schizophr Res. 2010 Nov;123(2-3):273-5. doi: 10.1016/j.schres.2010.07.016. Epub 2010 Aug 4. No abstract available. PMID 20688481